CLINICAL TRIAL: NCT04688827
Title: Impact of Different Types of Resistance Training Additional to Endurance Training During Rehabilitation Therapy in Patients With Heart Failure
Brief Title: Impact of Additional Resistance Training During Rehabilitation Therapy in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020044
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: heart failure; resistance training; rehabilitation therapy
MeSH Terms: conditions — Heart Failure | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group 1: low-intensity resistance training (Experimental)
  Interventions: Other: Exercise therapy
- training group 2: moderate-intensity resistance training (Experimental)
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — 15 weeks of resistance training (additional to endurance training)

SUMMARY:
The impact of moderate- or low-intensity resistance training will be investigated additional to endurance training in heart failure patients following rehabilitation. The aim is to optimize intensity of resistance training in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure and participation in cardiac rehabilitation

Exclusion Criteria:

* Orthopedic disorders, neurological disorders affecting muscle strength, cognitive disorders, heart or arterial surgery (percutaneous coronary intervention, bypass, heart valve surgery) in the last year, acute myocardial infarction in the last 6 months, participation in another intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
VO2peak | Prior to the intervention
  Maximal oxygen consumption during cardiopulmonary exercise test
VO2peak | After 15 weeks of intervention
  Maximal oxygen consumption during cardiopulmonary exercise test
VO2peak | After 24 weeks of follow-up
  Maximal oxygen consumption during cardiopulmonary exercise test

SECONDARY OUTCOMES:
Muscle strength | Prior to the intervention
  One-repetition maximum test (1RM) to evaluate maximal contraction of the muscle
Muscle strength | After 15 weeks of intervention
  One-repetition maximum test (1RM) to evaluate maximal contraction of the muscle
Muscle strength | After 24 weeks of follow-up
  One-repetition maximum test (1RM) to evaluate maximal contraction of the muscle
Functional capacity | Prior to the intervention
  Functional capacity evaluated via the six-minute walking test
Functional capacity | After 15 weeks of intervention
  Functional capacity evaluated via the six-minute walking test
Functional capacity | After 24 weeks of follow-up
  Functional capacity evaluated via the six-minute walking test
Quality of life in heart failure patients | Prior to the intervention
  Evaluation via Minnesota living with heart failure questionnaire
Quality of life in heart failure patients | After 15 weeks of intervention
  Evaluation via Minnesota living with heart failure questionnaire
Quality of life in heart failure patients | After 24 weeks of follow-up
  Evaluation via Minnesota living with heart failure questionnaire
Cardiac function | Prior to the intervention
  left-ventricular ejection fraction evaluated by transthoracic echocardiography
Cardiac function | After 15 weeks of intervention
  left-ventricular ejection fraction evaluated by transthoracic echocardiography
Cardiac function | After 24 weeks of follow-up
  left-ventricular ejection fraction evaluated by transthoracic echocardiography
Anthropometric measurements | Prior to the intervention
  body weight evaluated to determine body mass index
Anthropometric measurements | After 15 weeks of intervention
  body weight evaluated to determine body mass index
Anthropometric measurements | After 24 weeks of follow-up
  body weight evaluated to determine body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium